## **Informed Consent** · Informed Notification Page

Protocol Name: Correlation between Sphingolipid Metabolites and Liver

Failure after Hepatectomy

Solution Version Number: 1st Edition

Informed Consent Version and Date: 2<sup>nd</sup> Edition November 20, 2019 Research Institution: Southern Hospital of Southern Medical University

Lead Researcher: Zhou Jie

## Dear patient:

You will be invited to participate in a clinical study. This informed consent form provides you with information to help you decide whether to participate in this clinical study. Please read it carefully. If you have any questions, please ask the researcher responsible for the research.

Your participation in this study is voluntary. This research has been reviewed by the ethics review committee of this research institution.

- (1) Research Background and Research Purposes: Sphingolipid metabolites are significantly associated with the development of various liver diseases. The liver is an important organ of sphingolipid metabolism. We believe that the occurrence and development of liver failure after hepatectomy may have abnormal levels of sphingolipid metabolites. This subject will quantitatively and qualitatively analyze plasma and liver tissue sphingolipid metabolites in patients with hepatectomy, and collect perioperative clinical data to study the correlation between sphingolipid metabolites and liver failure after hepatectomy, and explore sphingolipid metabolites. The clinical significance of horizontal diagnosis and treatment of liver failure after hepatectomy.
- (2) Research Process: If you agree to participate in the study, we will number each subject, remove any characters that identify you, and create a medical record file. During the course of the study, we need to collect some of your specimens, including blood specimens and surgically removed abandoned liver tissue, during your routine clinical treatment. The time of collection includes blood collection before surgery, and early morning after surgery. Excised liver tissue is collected in blood and surgery. By health care

- professionals for your sampling, blood collection by additional nurses drawn routine from the arm when your blood clinical blood 5ml, 2 times: abandoned after liver tissue will totaling take 50- 100 mg surgeon. The blood collection time of this study is consistent with the medical-related blood collection time, without increasing the number of blood collections during your hospital stay. Your sample is for this study only.
- (3) Risk and Discomfort: Your sample collection will be performed strictly in accordance with the sterility requirements and will be performed during routine clinical blood draw without increasing the number of blood collections during your hospital stay. Medical blood collection may have some very small risks, including short-term pain, local bruising, a few people with mild dizziness, or extremely rare needle infections. If such a situation occurs, it will be treated according to the corresponding medical principles.
- (4) Benefits: Testing your specimens will help advance the diagnosis of the disease, may provide the necessary advice for your treatment, or provide useful information for the study of the disease, or may not.
- (5) Relevant Fees: You do not need to pay research fees for this study.
- (6) If you participate in the study, you will need to do the following: We will collect the clinical examination data during your stay and will save it for a long time after removing any characters that have an identification effect on your identity.
- (7) Privacy Issues: If you decide to participate in this study, your participation in the trial and the personal data in the trial are confidential. Your specimen will be identified by the research number number instead of your name. Other information that identifies you will also be identified unless you have your permission. All research members and research sponsors are required to keep your identity confidential. Your files will be kept in a locked filing cabinet for researcher only. To ensure that research conducted in accordance with the if of the regulations, necessary, а member government administration or institutional review board can review your personal information in accordance with the provisions research unit. When the results of this study are published, you will not disclose any of your personal information.
- (8) Damage Compensation: This study is a non-intervention study and in principle will not cause damage to your health. If damage to your health is caused, the Southern Hospital of Southern Medical University will provide compensation according to law.
- (9) How can I get more information?

You can ask any questions about this research at any time. Your doctor will leave you his / her phone number to answer your questions. Your doctor will promptly notify you if there is any important new information during the study that may affect your willingness to continue your research.

(10) Can voluntarily choose to participate in research and drop out of research

Whether or not to participate in the study is entirely up to your willingness. You may decline to participate in the study or withdraw from the study at any time during the study, which will not affect your relationship with the doctor and will not affect your medical or other benefits. Your doctor or researcher may discontinue your participation in this study at any time for your best interest.

## (11) What should I do now?

It is up to you to decide whether to participate in this study. You can discuss it with your family or friends before making a decision. Before you make a decision to participate in the study, please ask your doctor as much as possible until you fully understand the study. Thank you for reading the above materials. If you decide to participate in this study, please tell your doctor that he / she will arrange all the research for you. Please keep this information.

## **Informed Consent** · Signature Notification Page

I have read this informed consent form.

I have a chance to ask questions and all questions have been answered.

I understand that participation in this study is voluntary.

I will receive a copy of the signed Informed Consent Form.

I may choose not to participate in this study, or to withdraw from the researcher at any time without discrimination or retaliation, and my medical treatment and benefits will not be affected.

If I need other treatments, or if I don't follow the research plan, or if there is a research-related injury or any other reason, the researcher can stop me from continuing to participate in the study.

| Subject Name: |
|---|
| Subject signature: |
| Date: |
| Subject legal agent signaturedate: |
| (if applicable) |
| Contact number: |
| ( Note: If the subject is illiterate, the witness needs to be signed by the |
| witness, and if the subject is incapacitated, the agent must sign it ) |
| I have accurately informed the subject that he/she has accurately read this |
| informed consent and that the subject has an opportunity to ask a question. I |
| certify that he/she is willing to do so. |
| Researcher Name: |
| Researcher's Signature: |
| Date: |
| Contact number: |